CLINICAL TRIAL: NCT02398266
Title: Contrast Ultrasound Perfusion Imaging in PAD With Sonazoid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Sonazoid in PAD
Record Dates: First submitted 2015-03-03; First posted 2015-03-25 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy subjects (Experimental): Intervention: administration of ultrasound contrast agent (drug) to assess muscle perfusion. Normal healthy subjects (n=10) will be used for optimization of dose and acoustic settings for performing real-time contrast ultrasound perfusion imaging of the limb.
  Interventions: Drug: Contrast ultrasound of leg muscle with Sonazoid (Contrast ultrasound microvascular perfusion imaging)
- Patients with PAD and ABI 0.4-0.6 (Experimental): Intervention: administration of ultrasound contrast agent (drug) to assess muscle perfusion. Patients with moderate to severe PAD (ABI 0.4 to 0.6) will be evaluated with contrast ultrasound perfusion imaging using methods optimized in the first Arm to determine whether symptoms better correlate with perfusion imaging than other measures of PAD severity.
  Interventions: Drug: Contrast ultrasound of leg muscle with Sonazoid (Contrast ultrasound microvascular perfusion imaging)
- Patients with PAD Undergoing Revascularization (Experimental): Intervention: administration of ultrasound contrast agent (drug) to assess change in muscle perfusion produced by revascularization (surgical or percutaneous procedure). Patients with symptomatic PAD will be evaluated with contrast ultrasound perfusion imaging using methods optimized in the first Arm before and within 1 month of revascularization to determine whether improvement in symptoms correlate with perfusion imaging data.
  Interventions: Drug: Contrast ultrasound of leg muscle with Sonazoid (Contrast ultrasound microvascular perfusion imaging)

INTERVENTIONS:
Drug: Contrast ultrasound of leg muscle with Sonazoid (Contrast ultrasound microvascular perfusion imaging) — Skeletal muscle perfusion assessment of the thigh and calf skeletal muscle will be performed with contrast ultrasound of leg muscle with Sonazoid while at rest and during exercise stress
  Other Names: Contrast ultrasound microvascular perfusion imaging; Sonazoid

SUMMARY:
The measurement of limb skeletal muscle perfusion and perfusion reserve during exercise is an approach that can assess the total impact of the complex pathophysiologic processes in patients with limb ischemia, particularly in those with diabetes in whom distal arterial disease and abnormal microvascular functional responses are common. This trial is designed to: (a) optimize methods for assessment of limb perfusion at rest and during stress using contrast-enhanced ultrasound (normal subjects) and a microbubble contrast agent that is able to provide non-linear signal without destruction at medium acoustic pressures, and (b) to test whether perfusion imaging provides incremental information on the severity of disease in patients with peripheral artery disease.

ELIGIBILITY:
Inclusion Criteria:

* For Healthy controls: no active major medical problems or vasoactive medications
* For PAD: Known diagnosis with PAD an ABI of 0.4-0.6

Exclusion Criteria:

* Rutherford class 6 or greater
* Allergy to ultrasound contrast agents
* Previous limb amputation
* Pregnancy
* Known congenital or acquired right to left shunt

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle perfusion as measured by contrast ultrasound with Sonazoid microbubbles | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States